CLINICAL TRIAL: NCT07228962
Title: Using a Non-invasive Micro-suction Biomarker Extraction Device to Understand Atopic Eczema in Babies
Brief Title: Cutaneous Biomarkers in Atopic Eczema Using a Non-Invasive Micro-Suction Device in Babies
Acronym: CARE
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Engineering and Physical Sciences Research Council, UK (Other)
Responsible Party: Sponsor
Other Study IDs: 173024; EP/X013251/1 (Other Grant/Funding Number: Engineering & Physical Sciences Research Council)
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Eczema; Atopic Dermatitis; Atopic Eczema
Keywords: Eczema; Atopic Dermatitis; Immune System; Skin Barrier; Dermatology; Interstitial Skin Fluid; Microbiome; Early life
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Skin ISF samples - for immune marker, cytokine and metabolite analysis Skin Swabs - for skin microbiome and metabolome analysis
  These samples will be stored until all analysis for this study is complete before being disposed of in accordance with national Research Governance guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy babies: Babies up to 6 months old without eczema
- Babies with Eczema: Babies up to 6 months old with eczema

SUMMARY:
This project aims to establish whether an adapted extraction device is tolerable and will be able to measure chemical signals in baby's ISF. Insight into the chemical profiles found in the skin interstitial fluid (ISF) of healthy and diseased babies will identify signals that can be used to investigate the causes of eczema and propose new preventative strategies and effective treatments.

Specifically, it aims to:

1. Demonstrate that the developed ISF device can be used to extract biomarkers from the skin of babies non-invasively and is tolerable (not causing significant discomfort, bruising, or blister formation).
2. Compare the profile of chemical markers present in the ISF of healthy babies with babies that have developed eczema.
3. Compare the biomarker levels extracted from babies with eczema in lesional and non-lesional skin using the developed ISF device.
4. Compare the microbiome and metabolome profiles from swabs taken from babies with healthy skin and with eczema in lesional and non-lesional skin (exploratory outcome).

DETAILED DESCRIPTION:
Eczema is a skin condition that affects up to 20% of children worldwide, and its numbers are increasing. Our goal is to learn more about eczema by studying how immune signals in the skin differ between babies with eczema and those with healthy skin. To do this, investigators will gently use a non-invasive device to extract a tiny amount of fluid from the top layer of baby's skin(Interstitial Skin Fluid). By studying these samples, investigators want to compare the immune signals of healthy skin and skin affected by eczema. This research aims to deepen our understanding of why eczema causes inflammation and to identify the specific signals involved in this process, particularly in babies.

A total of 30 babies will be recruited, of which 15 will be healthy and 15 have eczema. They will be invited to attend for one visit lasting 1-1.5 hours. During the study visit, clinical information such as demographics, medical history and co-morbidities as well as eczema treatments (where applicable) and other skin care practices will be collected. For babies that have eczema, an eczema area and severity index (EASI) assessment will be conducted. For all participants enrolled onto the study, Interstitial Skin Fluid (ISF) samples will be extracted from the skin using a painless, non-invasive device that is well-tolerated and will not cause any pain or skin damage to the baby. Samples for assessing the skin microbiome will be collected, including skin swabs and tape strips taken in a pain-free manner. Skin barrier function assessments such as Transepidermal water loss (TEWL) will also be performed helping us understand how well the baby's skin holds onto moisture. This is a painless and non-invasive device that doesn't cause any discomfort to the baby.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy babies and babies with atopic dermatitis up to 6 months old.
2. Ability of parents/guardians/caregivers to provide written informed consent for study participation.
3. Willingness of parents/guardians/caregivers to comply with all study requirements.
4. Parents/guardians/caregivers competent use of English language.

Exclusion Criteria:

1. Parents/guardians/caregivers unable to give informed consent.
2. Preterm birth (defined as birth before 37 completed weeks gestation).
3. Significant inflammatory skin disease at birth.
4. Baby has any other serious health issue.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Babies up to 6 months old with or without eczema that can attend St Thomas' Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Cytokine levels in ISF | At enrolment
  The ISF extraction device will be applied to the baby's calf for a total of 5 min (both lesioned and non-lesioned skin in eczema presenting babies) and an ISF sample will be collected using an extraction gauze. The amount of protein or sodium will be used to determine the volume of ISF sampled. In addition, the release of soluble mediators such as IL-10 and TGF-beta as well as other Th1/Th2 cytokines IFN-Ɣ IL-1β IL-2 IL-4 IL-5 IL-13 IL-6 IL-8 (CXCL8) IL-10, IL-33, IL-12p70, TNF-α, GM-CSF, TSLP will be measured using an MSD cytokine analyser.

SECONDARY OUTCOMES:
TEWL | At enrolment
  TEWL, a validated measure of skin barrier function, will be measured using a closed chamber TEWL instrument (Biox Aquaflux Model AF200) near the ISF sampling site.
Microbiome profiles and Metabolite levels | At enrolment
  Microbiome and metabolome swabs will be taken, in healthy babies just from one site, in those with eczema from both lesional and non-lesional skin.
Tolerability of the use of the ISF Device | At enrolment
  Tolerability of the use of the non-invasive ISF device in babies with and without eczema will be assessed through a 5-point scale by the study team member, where score 1= very good; 2= good; 3= acceptable; 4= poor and 5= very poor. Photographs will be taken to record the observations. We will also measure tolerability quantitatively by measuring TEWL immediately after application of the device.
Investigator Assessments | At enrolment
  Changes in the skin will be observed and recorded by the investigator, including the Eczema Area and Severity Index (EASI) scoring, on a scale of 0-72, where a higher score corresponds to more severe eczema.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Flohr, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Undecided